CLINICAL TRIAL: NCT03190889
Title: Neuromuscular Intervention Targeted to Mechanisms of ACL Load in Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Aaron Krych, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-001833; R01AR055563 (NIH)
Record Dates: First submitted 2017-05-15; First posted 2017-06-19 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Rehabilitation; ACL Reconstruction
Keywords: ACL Reconstruction; Rehabilitation; Sports Injury; Neuromuscular Intervention; Knee Injury
MeSH Terms: conditions — Athletic Injuries; Knee Injuries

STUDY DESIGN:
Intervention Model Description: Overall Strategy. This is a prospective, randomized, repeated measures single- blind clinical trial. The purposes of this study are to 1) stratify patient risk for second ACL injury, and 2) determine the effects of differential treatment intervention, including targeted neuromuscular training (TNMT), home program only (HOME) and standard clinical (STAN) training, on clinical, biomechanical, and neuromuscular performance measures associated with an increased ACL injury risk. After the initial ACL injury and study enrollment, all patients will participate in standardized pre-operative rehabilitation. They will then undergo surgery by a fellowship-trained sports medicine surgeon at Mayo Clinic, Rochester, MN. Data for Aim 1 will be obtained from biomechanical, neuromuscular and clinical testing performed during Pre-Testing. Data for Aim 2 and the Exploratory Aim will be obtained from biomechanical and clinical test results obtained from Pre- and Post-Testing time points.
Who Masked: Participant, Investigator
Masking Description: Subjects are masked from group assignment. Group assignment is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care Group (No Intervention): Patients in the STAN group will participate in twelve sessions of supervised physical therapy over a six week period. Patients will participate in agility and plyometric drills, and continue strength exercises from the previous treatment phase. The clinic program will be performed in conjunction with a home running program. Patients in this group will not receive feedback from the therapist regarding movement quality during activities.
- Control Group (Other): HOME Program is distinguished by patients participating in a home only intervention that consists of running and strengthening exercises performed twice a week for six weeks. No plyometric or agility drills are performed in this study arm. This represents the minimal intervention to prepare for a return to sports. No neuromuscular training or movement training beyond the sagittal plane will be performed.
  Interventions: Other: HOME
- Intervention Group with Neuromuscular Training (Experimental): Patients who are enrolled in the TNMT group will participate in 12 sessions of supervised outpatient physical therapy over a six week period. The TNMT protocol is distinguished by performance of exercises designed to enhance core and hip strength, performance of neuromuscular training exercise that are designed to correct movement flaws associated with second ACL injury25, providing verbal and visual feedback and performance of single leg drills on both legs.
  Interventions: Other: TNMT

INTERVENTIONS:
Other: HOME — At home rehabilitation following ACL reconstructive surgery as described in the HOME arm.
  Arms: Control Group
Other: TNMT — Standard of care, clinical rehabilitation following ACL reconstructive surgery with the addition of specified targeted neuromuscular training as described in the TNMT arm.
  Arms: Intervention Group with Neuromuscular Training

SUMMARY:
The overall goal of this project is to reduce risk of second anterior cruciate ligament (ACL) injury in vulnerable populations (active athletes between 14 = 24 years old) through the identification of relative injury risk groups based on subject-specific movement patterns prior to second injury, as well as through the determination of effect for differential rehabilitation protocols following initial ACL reconstruction and prior to return to sport. As nearly one-third of athletes who have a primary ACL injury and return to sport will experience a secondary injury, results from the proposed work will allow us to prospectively identify high risk patients who are the most appropriate recipients of enhanced treatment, including targeted training, which may reduce the risk of second ACL injury. Secondary ACL injury has the potential to end athletic careers, promote the development of osteoarthritis, and have debilitating effects on quality of life. Hence, the information gathered in this investigation will offer ACL injured athletes the optimal potential to reduce or potentially prevent these negative health effects before they are initiated.

DETAILED DESCRIPTION:
Importance of the problem. Second ACL injury, whether it is an insult to the ipsilateral graft or the contralateral ligament, is a growing problem after reconstruction. Besides missing an additional year of athletic participation, increasing health care costs, and increased psychological distress, re-injury and subsequent revision surgery have significantly worse outcomes compared with those after initial reconstruction. Second injuries have been reported to occur at a rate of 1 of 17 (6%) within the first two years of surgery. However, a second tear prevalence of 29% has been reported. This is substantially higher than initial ACL injuries, reported to occur at a rate of 1 in 60 to 100. Risk factors for second injury include younger athletes 6 who return to high-level sporting activities early. Both sexes are at risk for second ACL injury, with women reported as having higher risk of contralateral injury, and men having an increased risk of ipsilateral injury. Thus, it is critical to include both sexes in second ACL injury prevention programs.

Improvement in scientific knowledge and clinical practice: Patients have differential responses after ACL injury, including their functional abilities, movement biomechanics, neuromuscular performance, and quadriceps strength. Building from our prior funded work, the investigators propose to prospectively evaluate these varying patient characteristics in an attempt to identify distinct groups with differing levels of risk for second injury (Aim 1). Our previous work revealed that there were three risk groups among uninjured female athletes. The significance of identification of patient groups with distinct needs is profound. Prospective identification of at-risk patients who are the most appropriate recipients of enhanced treatment will likely reduce second ACL risk, and yield a more efficacious delivery of health care resources after ACLR. The Cincinnati group described this differentiation in ACL deficient patients as the 'rule of thirds,' with one third of patients able to function without limitations and not needing to undergo surgical stabilization, one third adapting their activity level without surgery, and one third requiring surgery to perform daily activities without knee instability. A classification scheme described by the University of Delaware also differentiates ACL deficient patients into groups of thirds including copers (no limit in abilities), non-copers (unable to function without knee instability) or potential copers (individuals who have the potential to function without ACLR). There is evidence these differences in functional abilities and movement characteristics persist after ACLR. A randomized clinical trial concluded individuals who exhibit poor knee stability and function after injury may require additional time to return to pre-injury functional levels. In addition, some may be unable to develop appropriate quadriceps strength symmetry to support a return to high-level sports. These data indicate not all patients experience the same magnitude or duration of impairments and symptoms after ACLR. Consequently, multiple post-operative rehabilitation strategies may be necessary to facilitate optimum patient care and outcomes.

Working from the rule of one-thirds, identification of distinct patient groups with unique needs after surgery is a novel approach for integration of optimum second injury prevention strategies. Primary-injury risk factors provide an important window into the underlying biomechanical and neuromuscular deficits that may persist after ACL injury and reconstruction. Using a statistical analysis clustering technique, distinct groups with relative risk for first-time ACL injury have been identified, including low, moderate and high risk groups. Single limb postural stability combined with biomechanical variables including vertical ground reaction force (vGRF), frontal plane hip adduction moment minimum, and pelvis angle during drop jump landings were identified as significant contributors to frontal plane knee loading, a surrogate for ACL injury risk. This work has demonstrated the existence of discernable groups of athletes that are more appropriate for targeted neuromuscular training (TNMT) intervention to prevent first-time ACL injury.

Factors that contribute to primary ACL injury risk provide an important window into the underlying deficits that may persist after ACL injury and reconstruction. Age and activity level are significant factors, as young active individuals are the most likely cohort to sustain a second ACL rupture. Surgical factors include decreased graft size, use of allograft tissue, vertical graft position, and a lax graft. Anatomical risk factors may also contribute to ACL injury risk and include an increase in the posterior-inferior lateral tibial plateau slope and decreased notch width. Genetic factors also likely play a role. While it is encouraging that so many potential factors have been identified which may contribute to second ACL injury risk, none of these factors can be modified through non-surgical intervention. Modifiable biomechanical and neuromuscular measures associated with second ACL injury have been identified. Previous work by our laboratory included a prospective clinical trial, athletes who had undergone ACLR underwent testing before a return to pivoting and cutting sports. Thirteen athletes sustained a subsequent injury. Specific injury predictive parameters identified during testing included a net internal rotation moment of the uninvolved hip, an increase in total frontal plane knee movement, greater asymmetry in internal knee extensor moment at initial contact, and deficits in single-leg postural stability of the involved limb. These parameters predicted second injury in this population with excellent sensitivity (0.92) and specificity (0.88).

Differences in functional abilities after ACLR may be differentiated by more than biomechanical and neuromuscular characteristics. Clinically measured muscle weakness may persist for years after ACLR. Quadriceps strength is strongly related to measurements of knee function in athletes who have undergone ACLR. While hamstrings strength alone may not show a significant effect on knee function following ACL injury and reconstruction, hamstrings activation may be an important component in neuromuscular control of the reconstructed knee, especially in females, who tend to be 'quadriceps dominant'. In addition, deficits in the hamstrings-quadriceps torque production ratio also appear to be a key variable in the primary ACL injury risk model. The relationship between muscle weakness and differential risk for second injury has not been established. An understanding of the interplay may, however, be critical to the development of effective, group-specific intervention programs and reduction of second-injury risk.

It is currently unknown if biomechanical and clinical measures may effectively discern groups of patients who are at greatest risk for second ACL injury. Evaluation of movement mechanics and clinical characteristics, including strength, limb stability and self-reported function, at the time a patient initiates sports-specific training may yield insight to differential responses after ACLR. If distinct patient groups are identified, this information may be used to provide differentiated interventions based on risk for second injury. In Aim 2 of this proposal, the investigators will evaluate the effects of differential rehabilitation interventions. Our Exploratory Aim will be the initial step in translating the biomechanics-based, group algorithm into a clinical application for individualized categorization of risk. The results of this work may instigate a paradigm shift in treatment, and promote a more efficacious utilization of healthcare resources by providing enhanced care to those patients who are at greatest risk for secondary injury.

Impact on patient care. One of the factors that contributes to second ACL injury is incomplete or ineffective rehabilitation. Aberrant neuromuscular and biomechanical patterns are commonly seen up to 2 years after ACLR and may help explain the high rate of second ACL injury. Deficits in the neuromuscular control of both lower extremities following ACLR have been directly implicated in the risk for second ACL injury and may not only be a result of the initial knee injury and subsequent surgery, but may also characterize the athlete's pre-injury movement patterns. Therefore, identification and subsequent targeted treatment of aberrant post-ACLR movement patterns for both limbs are critical not only to maximize functional recovery but also to reduce the risk for second ACL injury. Though neuromuscular training programs result in a 73.4% decreased risk of a non-contact primary-ACL injury compared to those who do not participate in neuromuscular training, the efficacy of similar programs for reduction of second-ACL injury risk has not been examined.

An evidence-based targeted neuromuscular training (TNMT) program has been designed to prevent second ACL injury. This training program was developed with consideration to modifiable factors related to second-injury risk, the principles of motor learning, and careful selection of the exercises that may most effectively modify aberrant neuromuscular programs. In Aims 2 and 3 of this competing renewal proposal the investigators will evaluate the effects of differential treatment interventions. Notably, the investigators will assess the effectiveness of TNMT, including the utilization of visual and verbal biofeedback. Validation of this evidence-based, late-phase TNMT program may significantly impact clinical practice patterns through its integration in rehabilitation settings, and serve as a critical factor in reduction of second injury risk. Ultimately, determining if less intensive HOME and STAN training programs are effective interventions for patients who are at reduced risk for second ACL injury may prove to be a tremendous time and cost savings for patients and the health-care system.

ELIGIBILITY:
Inclusion Criteria:

* Age, 13 ≥ 30 years
* Acute (< 6 months), first-time, isolated ACL injury
* No history of previous knee surgery to either extremity
* No low back or lower extremity injury in the year prior to ACL injury necessitating medical care
* Pre-injury participation in cutting, jumping or pivoting sports for ≥ 50 hours/year
* Mechanism of injury did not involve a direct blow to the knee.
* Patients who sustain a medial collateral ligament (MCL) injury are eligible for study participation if medial knee instability is resolved prior to surgery
* Patients with simple meniscus tears (i.e., 2 cm vertical longitudinal tear) that do not necessitate alterations in rehabilitation will be eligible for study participation

Exclusion Criteria:

* History of previous knee surgery to either extremity
* Low back or lower extremity injury in the year prior to ACL injury necessitating medical care
* Second or greater ACL injury
* Greater than 6 months since occurrence of ACL injury
* Lack of participation in cutting, jumping, or pivoting sport
* Mechanisms of injury involved a direct blow of force to the knee
* Patients with MCL injury that exhibits unresolved medial knee instability
* Patients with complex, repairable meniscus tears (i.e., radial or root repair) and patients with full thickness articular cartilage lesions will not be eligible for participation secondary to significant alterations to postoperative rehabilitation protocol

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Planned distribution of subjects: US census reports for 2014 indicate the female sex comprises approximately 50% of the population in Olmsted (Rochester, MN) county. We therefore anticipate women will comprise approximately half of the study population.
Enrollment: 150 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Krych, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Emory University, Flowery Branch, Georgia
  - Mayo Clinic Square, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects over 1 hour drive (50 miles) away from the treatment facility were limited to STAN or HOME group randomization.
Groups:
- STAN: Patients in the STAN group will participate in twelve sessions of supervised physical therapy over a six week period. Patients will participate in agility and plyometric drills, and continue strength exercises from the previous treatment phase. The clinic program will be performed in conjunction with a home running program. Patients in this group will not receive feedback from the therapist regarding movement quality during activities.
- HOME: HOME Program is distinguished by patients participating in a home only intervention that consists of running and strengthening exercises performed twice a week for six weeks. No plyometric or agility drills are performed in this study arm. This represents the minimal intervention to prepare for a return to sports. No neuromuscular training or movement training beyond the sagittal plane will be performed.
  HOME: At home rehabilitation following ACL reconstructive surgery as described in the HOME arm.
- TNMT: Patients who are enrolled in the TNMT group will participate in 12 sessions of supervised outpatient physical therapy over a six week period. The TNMT protocol is distinguished by performance of exercises designed to enhance core and hip strength, performance of neuromuscular training exercise that are designed to correct movement flaws associated with second ACL injury25, providing verbal and visual feedback and performance of single leg drills on both legs.
  TNMT: Standard of care, clinical rehabilitation following ACL reconstructive surgery with the addition of specified targeted neuromuscular training as described in the TNMT arm.
Period: Overall Study
Arm/Group | STAN | HOME | TNMT
Started | 51 | 50 | 49
Completed | 38 | 33 | 42
Not Completed | 13 | 17 | 7
Not completed — Lost to Follow-up | 7 | 7 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Did not complete protocol | 4 | 9 | 0
Not completed — COVID-19 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Subjects who consented, but never showed up for the pretesting analysis session were excluded. This included two (2) STAN, two (2) HOME, and two (2) TNMT subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | STAN | HOME | TNMT | Total
Number analyzed (Participants) | 49 | 48 | 47 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 31 | 35 | 102
  Between 18 and 65 years | 13 | 17 | 12 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.90 (3.03) | 18.19 (4.11) | 16.98 (3.19) | 17.35 (3.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 32 | 84
  Male | 23 | 22 | 15 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 46 | 45 | 46 | 137
  Unknown or Not Reported | 1 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 6 | 21
  White | 37 | 35 | 38 | 110
  More than one race | 4 | 2 | 2 | 8
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 47 | 144
Height [Mean (Standard Deviation); unit: centimeters] | 170 (11) | 172 (8) | 169 (7) | 170 (9)
Mass [Mean (Standard Deviation); unit: kilograms] | 72.36 (15.66) | 68.93 (14.52) | 70.27 (18.20) | 70.52 (16.13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Second ACL Injury
Description: Subjects recruited for this investigation will be recovering from primary ACL injury. Participants will be monitored for injury history from time of enrollment in study. Report of any additional ACL injury whether contralateral leg or involved leg will be counted as a second ACL injury.
Time Frame: 12-48 months
Population: Only subjects who completed both pre and post-testing assessments and completed at least one year of subsequent injury tracking were included.
Measure: Count of Participants; unit: Participants
Arm/Group | STAN | HOME | TNMT
Number analyzed (Participants) | 27 | 28 | 32
Participants | 3 | 7 | 5

2. Secondary Outcome: Frontal Plane Knee Kinetics
Description: Joint moments at the knee will be recorded from study participants as they perform athletic tasks. Frontal plane knee moments have previously been associated with ACL injury risk and will be used to assess the proposed treatment groups.
Time Frame: Change after 6 weeks of interventional protocol
Reporting Status: Not Posted, anticipated posting 2025-08

3. Secondary Outcome: Frontal Plane Knee Kinematics
Description: Joint excursion and angles at the knee will be recorded from study participants as they perform athletic tasks. Frontal plane excursion and angle has been associated with increased frontal plane moments that are associated with increased relative risk of ACL injury.
Time Frame: Change after 6 weeks of interventional protocol
Reporting Status: Not Posted, anticipated posting 2025-08

ADVERSE EVENTS:
Time Frame: 12-48 months
Description: Record of adverse events occuring during interventional training sessions or during the pre- and post-intervention assessment sessions.
Arm/Group | STAN | HOME | TNMT
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03190889/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03190889/ICF_001.pdf